CLINICAL TRIAL: NCT06094036
Title: Physical Exercise as a Sustainability Tool in Men Affected With Metabolic Syndrome-related Late-onset Central Hypogonadism: Role of Endocrine-metabolic and Neurovegetative Outcomes
Brief Title: Physical Exercise as a Sustainability Tool in Men With Dysmetabolic Hypogonadism
Acronym: ExLOH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 45C202
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hypogonadism, Male; Metabolic Syndrome; Autonomic Imbalance; Life Style, Healthy; Physical Inactivity
MeSH Terms: conditions — Eunuchism; Metabolic Syndrome; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weekly physical activity volume performed above 600 MET·minutes/week (Other): Exercise program requiring clear definition of modality, intensity, frequency, duration and progression of exercise, tailored on patient's clinical conditions and goals.
  Interventions: Behavioral: Structured and personalized program of physical exercise
- weekly physical activity volume performed below 600 MET·minutes/week (Other): Exercise program requiring clear definition of modality, intensity, frequency, duration and progression of exercise, tailored on patient's clinical conditions and goals.
  Interventions: Behavioral: Structured and personalized program of physical exercise

INTERVENTIONS:
Behavioral: Structured and personalized program of physical exercise — In line with the most recent guidelines, exercise prescription will require the clear definition of modality, intensity, frequency, duration and progression of exercise, tailored on patient's clinical conditions and goals.
  This intervention will be accompanied by a nutrition program aiming for proper dietary habits in terms of both quantity and quality.

SUMMARY:
Aim of this project is to delineate sustainable physical exercise programs and to assess the effects of such programs mainly on endocrine-metabolic and neurovegetative outcomes in a cohort of men with metabolic syndrome-related late-onset central hypogonadism.

Participants will undergo a personalised exercise program. After 6 months they will be subdivided into two groups, according to the weekly physical activity volume actually performed (above or below 600 MET·minutes/week). Changes in endocrine-metabolic and neurovegetative outcomes will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of late-onset central hypogonadism: total T levels < 8 nmol/L (or < 12 nmol/L in the presence of calculated free T < 225 pmol/L) combined with sexual symptoms (erectile dysfunction, low libido and loss of waking erections) [12];
* diagnosis of metabolic syndrome, defined as association of waist circumference (WC) > 94 cm and at least two among the following criteria: triglycerides ≥ 150 mg/dl, HDL-C < 40 mg/dl, glucose > 100 mg/dl, blood pressure (BP) ≥ 130/85 mmHg [33];
* ability to give informed consent, in accordance with good clinical practice rules and applicable national laws.

Exclusion Criteria:

* History of hypothalamus-pituitary organic disorders and/or testicular diseases;
* impossibility to assess cardiac autonomic regulation due to arrhythmias and/or current treatment for heart rate (HR) control (e.g., beta-blockers, antiarrhythmics);
* impossibility to undergo clinical assessment;
* impossibility or contraindications to perform exercise program (for instance, psychiatric disorders, severe musculoskeletal diseases, arrhythmias);
* inability to give informed consent or unwillingness to be enrolled in the study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
change in hypothalamic-pituitary-gonadal axis function | 6 months
  particularly testosterone levels (nmol/l)

SECONDARY OUTCOMES:
Change in body composition | 6 months
  percentage of fat mass and free fat mass
Change in serum skeletal isoenzyme of alkaline phosphatase | 6 months
  Change in serum skeletal isoenzyme of alkaline phosphatase concentration (ug/l)
Change in C-terminal telopeptide of type I collagen | 6 months
  Change in C-terminal telopeptide of type I collagen concentration (ng/l)
Change in erythrocyte sedimentation rate | 6 months
  Change in erythrocyte sedimentation rate (mm/h)
Change in C-reactive protein | 6 months
  Change in C-reactive protein concentration (mg/l)
Change in total cholesterol | 6 months
  Change in total cholesterol concentration (mg/dl)
Change in HDL cholesterol | 6 months
  Change in HDL cholesterol concentration (mg/dl)
Change in triglycerides | 6 months
  Change in triglycerides concentration (mg/dl)
Change in glucose profile | 6 months
  glycemia (mg/dl)
Change in kidney function | 6 months
  creatinine (mg/dl)
Change in aspartate aminotransferase | 6 months
  Change in aspartate aminotransferase concentration (U/L)
Change in alanine aminotransferase | 6 months
  Change in alanine aminotransferase concentration (U/L)
Change in cardiac autonomic regulation | 6 months
  Autonomic Nervous System Index (ANSI)
Change in nutrition quality | 6 months
  American Heart Association (AHA) Diet Score
Change in perception of stress, fatigue, and somatic symptoms | 6 months
  short version of 4SQ questionnaire considering 4 specific symptoms (total score ranging from 0 to 40)
Change in weekly physical activity volume | 6 months
  short version of International Physical Activity Questionnaire, which focuses on intensity (nominally estimated in Metabolic Equivalents - MET - according to the type of activity) and duration (in minutes) of physical activity. The following levels will be considered: brisk walking (≈ 3.3 METs), other modalities of activity of moderate intensity (≈ 4.0 METs), and activities of vigorous intensity (≈ 8.0 METs).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Lucini, MD, PhD, Principal Investigator — University of Milan; Istituto Auxologico Italiano, IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy